CLINICAL TRIAL: NCT00000298
Title: Buprenorphine Combination Tablet Feasibility
Brief Title: Buprenorphine Combination Tablet Feasibility - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09260-1; P50-09260-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 1996-01

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

INTERVENTIONS:
Drug: Buprenorphine/naloxone

SUMMARY:
The purpose of this study is to determine target dose range of buprenorphine/naloxone combination tablet that provides therapeutic response in opiate addicts with low to moderate dependence, and to identify appropriate initial induction dose in opiate addicts with low to moderate dependence."

ELIGIBILITY:
Inclusion Criteria:

Males/Females ages 21-50, opiate dependence according to DSM-IV criteria, self-reported use within the last 30 days, agreeable to conditions of study and signed informed consent

Exclusion Criteria:

Psychiatric disorder that requires medication therapy, history of seizures, pregnant and/or nursing women, dependence on etoh or benzodiazepines or other sedative-hypnotics, acute hepatitis, other medical conditions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1995-08

PRIMARY OUTCOMES:
Withdrawal symptoms
Opiate use
Opiate craving

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States

REFERENCES:
- [Background] Buprenorphine/nalaxone cmbination tablet: First clinical experience (j. Add Dis 1997, in press). Buprenorphine/naloxone combination tablet: First clincial experience (J Add Dis 1997, in press).